CLINICAL TRIAL: NCT00460239
Title: Evaluation of Opioid Antagonist Activity in Humans
Brief Title: Buprenorphine's Dose Response Curve
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-08045-8; 5R01DA008045-08 (NIH); R01DA008045 (NIH); DPMCDA (Other: NIDA)
Record Dates: First submitted 2007-04-11; First posted 2007-04-13 (Estimated); Results first posted 2017-03-03 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Opioid-related Disorders
Keywords: Opioid addiction; Opioid dependence; Buprenorphine
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine; Morphine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Placebo (Experimental): All participants are randomly assigned to receive an order of the 8 study drugs/doses (placebo, 2 doses of morphine, 5 doses of buprenorphine).
  Interventions: Drug: Placebo
- Morphine 15 (Experimental): All participants are randomly assigned to receive an order of the 8 study drugs/doses (placebo, 2 doses of morphine, 5 doses of buprenorphine).
  Interventions: Drug: Morphine
- Morphine 30 (Experimental): All participants are randomly assigned to receive an order of the 8 study drugs/doses (placebo, 2 doses of morphine, 5 doses of buprenorphine).
  Interventions: Drug: Morphine
- Buprenorphine 8 (Experimental): All participants are randomly assigned to receive an order of the 8 study drugs/doses (placebo, 2 doses of morphine, 5 doses of buprenorphine).
  Interventions: Drug: Buprenorphine
- Buprenorphine 16 (Experimental): All participants are randomly assigned to receive an order of the 8 study drugs/doses (placebo, 2 doses of morphine, 5 doses of buprenorphine).
  Interventions: Drug: Buprenorphine
- Buprenorphine 32 (Experimental): All participants are randomly assigned to receive an order of the 8 study drugs/doses (placebo, 2 doses of morphine, 5 doses of buprenorphine).
  Interventions: Drug: Buprenorphine
- Buprenorphine 48 (Experimental): All participants are randomly assigned to receive an order of the 8 study drugs/doses (placebo, 2 doses of morphine, 5 doses of buprenorphine).
  Interventions: Drug: Buprenorphine
- Buprenorphine 60 (Experimental): All participants are randomly assigned to receive an order of the 8 study drugs/doses (placebo, 2 doses of morphine, 5 doses of buprenorphine).
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine — Intramuscular, doses (8, 16, 32, 48, 60 mg) are blind; administered up to 1-2 times per week.
  Arms: Buprenorphine 16; Buprenorphine 32; Buprenorphine 48; Buprenorphine 60; Buprenorphine 8
Drug: Morphine — Intramuscular; up to 1-2 times per week; doses (15, 30 mg) double blind
  Arms: Morphine 15; Morphine 30
Drug: Placebo — Intramuscular; double blind; once per week
  Arms: Placebo

SUMMARY:
This is a residential study that looks at the effects of buprenorphine in persons who abuse but are not dependent on opioids. Animal studies show that very high doses of buprenorphine produce less effects than mid-range doses. This suggests that buprenorphine can be a very safe medication. However, no studies in humans have tested higher doses in a similar way. The goal of this study is to show the effects of single doses of buprenorphine, across a range of doses, in persons who are not physically dependent on opioids (but do abuse opioids).

DETAILED DESCRIPTION:
Preclinical studies have demonstrated for a variety of measures that buprenorphine has a bell-shaped dose response curve. However, human studies with buprenorphine have not shown such an effect, although controlled studies have generally not tested higher acute doses of buprenorphine. Current clinical recommendations generally place an upper limit of daily buprenorphine dosing at 32 mg of sublingual tablets, although considerably higher acute doses have been administered to humans (primarily in clinical studies of less than daily dosing). Determining the relationship between higher doses of buprenorphine in humans and effects produced would be valuable; it would be scientifically interesting to demonstrate a bell-shaped curve in humans, and it would help guide clinical practice (for example, with respect to dosing, safety, and side effect considerations. The purpose of this study is to characterize the dose response curve for buprenorphine in humans, utilizing acute single doses of parenteral buprenorphine.

ELIGIBILITY:
Inclusion Criteria:

1. current opioid abuse but not physically dependent on opioids

Exclusion Criteria:

1. evidence of significant medical (e.g., insulin dependent diabetes) or psychiatric (e.g., schizophrenia) illness
2. anemia defined as a hematocrit less than 30%
3. females are required to provide a negative pregnancy test prior to study participation
4. baseline electrocardiogram (ECG) showing prolongation of the corrected QT interval (QTc)
5. current significant alcohol or sedative/hypnotic drug use
6. Forced expiratory volume at one second (FEV1) of less than 50% at the time of screening
7. applicants seeking treatment for their substance abuse will not be admitted to the study, and should be provided information about treatment services available

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2007-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric C Strain, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University (BPRU) Bayview Campus, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Condition 1: Participants receive single doses of intramuscular (IM) test drugs; there were 9 possible test drugs (placebo [P], 2 doses of morphine [M], 5 doses of buprenorphine [B]), with at least 3 days between IM injections. For this condition, the order of dosing was (numbers represent doses in mg): B8, B16, B32, B48, B60, M15, M30, P.
- Condition 2: Participants receive single doses of intramuscular (IM) test drugs; there were 9 possible test drugs (placebo [P], 2 doses of morphine [M], 5 doses of buprenorphine [B]), with at least 3 days between IM injections. For this condition, the order of dosing was (numbers represent doses in mg): B8, B16, B32, M15, B48, P, B60, M30.
- Condition 3: Participants receive single doses of intramuscular (IM) test drugs; there were 9 possible test drugs (placebo [P], 2 doses of morphine [M], 5 doses of buprenorphine [B]), with at least 3 days between IM injections. For this condition, the order of dosing was (numbers represent doses in mg): B8, B16, B32, B48, M30, B60, P, M15.
- Condition 4: Participants receive single doses of intramuscular (IM) test drugs; there were 9 possible test drugs (placebo [P], 2 doses of morphine [M], 5 doses of buprenorphine [B]), with at least 3 days between IM injections. For this condition, the order of dosing was (numbers represent doses in mg): B8, M15, B16, P, B32, M30, B48, B60.
- Condition 5: Participants receive single doses of intramuscular (IM) test drugs; there were 9 possible test drugs (placebo [P], 2 doses of morphine [M], 5 doses of buprenorphine [B]), with at least 3 days between IM injections. For this condition, the order of dosing was (numbers represent doses in mg): B8, B16, M30, B32, P, B48, M15, B60.
- Condition 6: Participants receive single doses of intramuscular (IM) test drugs; there were 9 possible test drugs (placebo [P], 2 doses of morphine [M], 5 doses of buprenorphine [B]), with at least 3 days between IM injections. For this condition, the order of dosing was (numbers represent doses in mg): M15, P, B8, M30, B16, B32, P, B48, B60.
- Condition 7: Participants receive single doses of intramuscular (IM) test drugs; there were 9 possible test drugs (placebo [P], 2 doses of morphine [M], 5 doses of buprenorphine [B]), with at least 3 days between IM injections. For this condition, the order of dosing was (numbers represent doses in mg): M30, B8, P, B16, M15, B32, B48, B60.
- Condition 8: Participants receive single doses of intramuscular (IM) test drugs; there were 9 possible test drugs (placebo [P], 2 doses of morphine [M], 5 doses of buprenorphine [B]), with at least 3 days between IM injections. For this condition, the order of dosing was (numbers represent doses in mg): P, M30, M15, B8, B16, B32, B48, B60.
- Condition 9: Participants receive single doses of intramuscular (IM) test drugs; there were 9 possible test drugs (placebo [P], 2 doses of morphine [M], 5 doses of buprenorphine [B]), with at least 3 days between IM injections. For this condition, the order of dosing was (numbers represent doses in mg): M15, B8, B16, B32, M30, P, B48, B60.
Period: Overall Study
Arm/Group | Condition 1 | Condition 2 | Condition 3 | Condition 4 | Condition 5 | Condition 6 | Condition 7 | Condition 8 | Condition 9
Started | 0 | 3 | 1 | 0 | 1 | 4 | 1 | 1 | 1
Completed | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All Study Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (6.48)
Gender [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Peak Change From Baseline in Drug Effect Assessed by Visual Analog Scale (VAS)
Description: Opioid agonist effects measured by peak change from baseline drug effect visual analog scale. Scores range from 0 (not all all) to 100 (extremely); higher scores indicate a stronger drug effect.
Time Frame: Each experimental test session (8 experimental test sessions assessed for up to 6-7 weeks)
Population: Subjects who completed all test conditions.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo 0 mg | Morphine 15 mg | Morphine 30 mg | Buprenorphine 8 mg | Buprenorphine 16 mg | Buprenorphine 32 mg | Buprenorphine 48 mg | Buprenorphine 60 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
units on a scale | 17.75 (22.41) | 27.25 (33.50) | 29.63 (43.29) | 58.25 (32.58) | 48.50 (41.19) | 40.25 (35.07) | 57.63 (40.41) | 41.63 (36.56)

2. Primary Outcome: Psychomotor/Cognitive Performance Effects Assessed by Digit Symbol Substitution Test (DSST)
Description: Digit Symbol Substitution Test (DSST) is a sub-test within the Wechsler Adult Intelligence Scale and is frequently used to assess psychomotor performance changes associated with drug effects. The higher the percent correct on this measure the better the performance.
Time Frame: Each experimental test session (8 experimental test sessions assessed for up to 6-7 weeks)
Measure: Mean (Standard Deviation); unit: percentage of correct answers
Arm/Group | Placebo 0 mg | Morphine 15 mg | Morphine 30 mg | Buprenorphine 8 mg | Buprenorphine 16 mg | Buprenorphine 32 mg | Buprenorphine 48 mg | Buprenorphine 60 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
percentage of correct answers | 94.03 (10.21) | 91.60 (16.55) | 89.44 (18.33) | 90.91 (10.35) | 86.60 (19.98) | 83.17 (24.80) | 85.86 (19.21) | 77.99 (27.57)

3. Primary Outcome: Psychomotor/Cognitive Performance Effects Assessed by Trails B
Description: The Trails B task specifically measures set shifting and executive functioning within the Trail-Making Test. Part B consists of 25 circles distributed over a sheet of paper. Participants are asked to connect the circles in an ascending pattern, alternating between numbers and letters (i.e., 1-A-2-B-3-C, etc.). Results are reported as the number of seconds required to complete the task; therefore, higher scores reveal greater impairment.
Time Frame: Each experimental test session (8 experimental test sessions assessed for up to 6-7 weeks)
Population: Subjects who completed all test conditions.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo 0 mg | Morphine 15 mg | Morphine 30 mg | Buprenorphine 8 mg | Buprenorphine 16 mg | Buprenorphine 32 mg | Buprenorphine 48 mg | Buprenorphine 60 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
minutes | 1.58 (0.84) | 1.51 (0.82) | 1.68 (1.15) | 1.57 (0.66) | 1.85 (1.39) | 1.42 (0.39) | 1.49 (0.53) | 1.46 (0.50)

4. Primary Outcome: Physiologic Effects as Assessed by Blood Pressure
Time Frame: Each experimental test session (8 experimental test sessions assessed for up to 6-7 weeks)
Population: Subjects who completed all test conditions.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo 0 mg | Morphine 15 mg | Morphine 30 mg | Buprenorphine 8 mg | Buprenorphine 16 mg | Buprenorphine 32 mg | Buprenorphine 48 mg | Buprenorphine 60 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
mmHg
  Systolic Blood Pressure | 114.11 (8.82) | 114.71 (10.34) | 119.21 (10.85) | 118.59 (15.15) | 111.42 (9.43) | 114.11 (14.84) | 119.18 (12.48) | 116.77 (11.90)
  Diastolic Blood Pressure | 63.85 (7.13) | 64.92 (8.18) | 66.72 (8.08) | 67.35 (7.62) | 61.82 (6.96) | 62.60 (9.33) | 65.73 (7.29) | 64.39 (7.02)

5. Primary Outcome: Physiologic Effects as Assessed by Heart Rate
Time Frame: Each experimental test session (8 experimental test sessions assessed for up to 6-7 weeks)
Population: Subjects who completed all test conditions.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo 0 mg | Morphine 15 mg | Morphine 30 mg | Buprenorphine 8 mg | Buprenorphine 16 mg | Buprenorphine 32 mg | Buprenorphine 48 mg | Buprenorphine 60 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
beats/min | 70.44 (7.56) | 70.56 (6.04) | 69.80 (8.19) | 71.22 (9.61) | 69.41 (8.19) | 66.44 (10.20) | 69.06 (6.86) | 67.51 (8.24)

6. Primary Outcome: Physiologic Effects as Assessed by Body Temperature
Time Frame: Each experimental test session (8 experimental test sessions assessed for up to 6-7 weeks)
Population: Subjects who completed all test conditions.
Measure: Mean (Standard Deviation); unit: Degrees Fahrenheit
Arm/Group | Placebo 0 mg | Morphine 15 mg | Morphine 30 mg | Buprenorphine 8 mg | Buprenorphine 16 mg | Buprenorphine 32 mg | Buprenorphine 48 mg | Buprenorphine 60 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
Degrees Fahrenheit | 85.99 (5.41) | 87.43 (4.82) | 89.20 (3.91) | 89.76 (4.30) | 90.33 (3.84) | 89.11 (4.12) | 90.22 (4.25) | 90.62 (4.44)

7. Primary Outcome: Physiologic Effects as Assessed by Oxygen Saturation
Time Frame: Each experimental test session (8 experimental test sessions assessed for up to 6-7 weeks)
Population: Subjects who completed all test conditions.
Measure: Mean (Standard Deviation); unit: percentage of saturated hemoglobin
Arm/Group | Placebo 0 mg | Morphine 15 mg | Morphine 30 mg | Buprenorphine 8 mg | Buprenorphine 16 mg | Buprenorphine 32 mg | Buprenorphine 48 mg | Buprenorphine 60 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
percentage of saturated hemoglobin | 97.81 (0.77) | 97.57 (.80) | 97.15 (0.84) | 96.94 (0.96) | 96.73 (1.07) | 96.37 (1.61) | 96.75 (1.30) | 96.49 (1.62)

8. Primary Outcome: Physiologic Effects as Assessed by Pupil Diameter
Time Frame: Each experimental test session (8 experimental test sessions assessed for up to 6-7 weeks)
Population: Subjects who completed all test conditions.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Placebo 0 mg | Morphine 15 mg | Morphine 30 mg | Buprenorphine 8 mg | Buprenorphine 16 mg | Buprenorphine 32 mg | Buprenorphine 48 mg | Buprenorphine 60 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
millimeters | 4.00 (1.31) | 3.33 (0.87) | 2.74 (0.83) | 2.87 (1.19) | 2.73 (0.84) | 2.63 (0.79) | 2.61 (1.02) | 2.64 (0.99)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during time participants resided on the residential unit (target period of 6-7 weeks).
Arm/Group | Placebo Intervention | Morphine Intervention | Buprenorphine Intervention
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No